CLINICAL TRIAL: NCT03299023
Title: The Effect of Tooth Position During Orthodontic Treatment on the Apnea/ Hypopnea Index (AHI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Harvard School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Dr. Shaima Tabari, Investigator, Harvard School of Dental Medicine
Other Study IDs: R8-1648
Record Dates: First submitted 2017-09-13; First posted 2017-10-02 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Obstructive Sleep Apnea; Orthodontic Tooth Movement; Apnea; Sleep Disordered Breathing
Keywords: Obstructive Sleep Apnea; Orthodontics; Tooth Movement; Medibyte; Apnea; Hypopnea; Sleep; Disturbed Breathing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medibyte Portable Monitor — Patients will be provided with the portable monitor in order to measure their apnea/hypopnea index.

SUMMARY:
The study design of this research project involves orthodontic patients registered at the Harvard School of Dental Medicine who are deemed eligible to undergo orthodontic treatment and who have been provided with sufficient information to make informed consent to join the sleep study. These patients will be provided with the Medibyte sleep monitor and instructed on the proper manner in which it should be set up and worn for the one night study period. This process will be carried out twice throughout the course of the study, once before any orthodontic appliance has been cemented and once after the required amount of tooth movement has been attained with the orthodontic appliance still in place.

The de-identified data from the Medibyte monitor will be downloaded using the Braebon software and analyzed.

DETAILED DESCRIPTION:
The study design of this research project involves recruiting orthodontic patients registered at the Harvard School of Dental Medicine who are deemed eligible to undergo orthodontic treatment and who have been provided with sufficient information to make informed consent to join the sleep study. The participants will be provided with the Medibyte sleep monitor and instructed on the proper manner in which it should be set up and worn for the one or two night study period. The purpose of the Medibyte monitor is solely to provide a calibrated value of AHI. The Medibyte monitor will not be utilized for investigations and/or treat, cure, mitigate a medical condition. This process will be carried out twice throughout the course of the study, once before any orthodontic appliance has been cemented and once after the required amount of tooth movement has been attained with the orthodontic appliance still in place.

The de-identified data from the Medibyte monitor will be downloaded using the Braebon software and analyzed providing a baseline value and post orthodontic movement AHI value. Additionally the patients arch width, length and other orthodontic measurements will also be taken both from their 3-D dental models and also their 2-D lateral cephalogram x-ray all of which are part of the routine orthodontic records (the x-rays will be taken regardless of the patients participation in the study since they are a required component of the orthodontic records taken at HSDM). The values obtained from the patients casts, lateral cephalogram and Medibyte AHI values will be analyzed both pre-orthodontic appliance cementation and also post tooth movement. The changes, if any, in the dental parameters as compared with the AHI values will allow the investigation of the orthodontic effects of expanding the maxilla, moving the front teeth either forwards or backwards which in effect cause changes to the airway and its effect on AHI values during sleep. In addition to the measurements taken intra-orally, surveys will also be undertaken to study any changes the patients may experience in their sleep and quality of life. If the Medibyte shows a severe reading for obstructive sleep apnea, these patients will then be referred to a sleep specialist for further more conclusive testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults/children undergoing orthodontic care at HSDM

Exclusion Criteria:

* Patients already begun orthodontic therapy
* Patients obtaining orthognathic surgery
* Patients with high index of care need- have hypercapnia, hypoventilation, allergies or nose blockages

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients already registered at the Harvard School of Dental Medicine department of Orthodontics. Informed consent will be obtained before the questionnaires and portable monitor will be provided.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-05-10 (Estimated); Study Completion 2019-06-10 (Estimated)

PRIMARY OUTCOMES:
Relationship between dental movements and AHI | 2 Year
  This outcome aims to measure any changes in the dental measurements such as arch length, arch perimeter, inter-canine and inter-molar changes on the AHI value.
Relationship between skeletal changes and AHI | 2 Year
  This outcome aims to measure any changes in the skeletal changes such as SNA, SNB, ANB etc. as measured by the lateral cephalogram and any changes in the AHI
Relationship between airway cephalometric changes and AHI | 2 Year
  This outcome aims to measure any changes in the airway cephalometric measurements such as the upper/middle/superior airway space etc. and the AHI

SECONDARY OUTCOMES:
Relationship between the changes in the reported quality of life measurements and the AHI | 2 Year
  This outcome aims to measure any changes in the reported quality of life measurements as measured by questionnaires such as conners, epworth, pediatric quality of life and pediatric sleep quesitonnaire and the AHI vale.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No